CLINICAL TRIAL: NCT00939640
Title: Effects of the Dietary Approaches to Stop Hypertension(DASH) Sodium-restricted Diet on Ventriculovascular Function in Heart Failure With Preserved Systolic Function
Brief Title: Effects of the Dietary Approaches to Stop Hypertension(DASH) Sodium-restricted Diet in Diastolic Heart Failure
Acronym: DASH-DHF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Scott L. Hummel, Assistant Professor, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HUM00025253
Record Dates: First submitted 2009-07-14; First posted 2009-07-15 (Estimated); Results first posted 2018-10-22 (Actual); Last update posted 2019-10-15 (Actual); Status verified 2019-10

CONDITIONS: Diastolic Heart Failure; Hypertensive Heart Disease
Keywords: Diet; Sodium; Hypertension; Potassium; Antioxidants; congestive heart failure; Heart failure with normal ejection fraction; Heart failure with preserved systolic function
MeSH Terms: conditions — Heart Failure, Diastolic; Hypertension; Heart Failure | interventions — Dietary Approaches To Stop Hypertension; Diet, Sodium-Restricted

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dietary intervention (Experimental): Diet patterned after the intervention in the DASH-Sodium trial (Sacks FM et al. New Engl J Med 2001;344(1):3-10). The diet includes higher quantities of fresh fruits and vegetables, whole grain products, and low-fat dairy products than the standard American diet. The target sodium content is 50 mmol per 2100 kcal, and the caloric content is intended to maintain body weight. The diet is designed, prepared, and packaged by research dietitians and all food and beverages are provided for study participants.
  Interventions: Behavioral: DASH/sodium-restricted diet (SRD)

INTERVENTIONS:
Behavioral: DASH/sodium-restricted diet (SRD) — Baseline diet will be assessed via Block Food Frequency Questionnaire, and 24-hour urinary sodium, potassium, and 8-isoprostanes will be measured. Subjects will then be assigned to 21 days of the DASH/SRD, with all food and beverages provided. Adherence will be assessed through a three-day food diary at the midpoint of the intervention, and at the end of the study urinary sodium, potassium, and 8-isoprostanes will again be measured.
  Other Names: DASH diet; sodium-restricted diet; low sodium diet; DASH-sodium

SUMMARY:
Heart failure with preserved systolic function (HF-PSF, or 'diastolic heart failure') accounts for half of hospitalizations for heart failure in patients over the age of 65. Most HF-PSF patients have systemic hypertension (HTN), and characteristic HTN-induced cardiovascular changes contribute to HF-PSF. However, it is unclear why most patients with HTN never develop HF-PSF or which specific aspects of HTN predispose to HF-PSF.

In the Dahl S rat, the primary animal model of HF-PSF, high dietary sodium intake suppresses the systemic renin-angiotensin-aldosterone system, but upregulates renal and cardiac renin-angiotensin-aldosterone system by inducing oxidative stress. In humans, the magnitude of blood pressure response to sodium ingestion and depletion can categorize subjects as "salt-resistant" and "salt-sensitive." Human salt sensitivity is associated with structural and loading conditions that increase the risk for HF-PSF, including HTN, ventricular hypertrophy and diastolic dysfunction, arterial stiffening, and increased plasma volume. High dietary sodium intake induces oxidative stress in salt-sensitive humans. In humans with HTN and normal ventricular systolic function that do not have heart failure, increased oxidative stress predicts impaired exercise capacity, ventricular hypertrophy, diastolic dysfunction, arterial stiffening, and vascular endothelial dysfunction. The investigators have proposed that "salt sensitivity" and the accompanying oxidative stress on the typical high-sodium Western diet may contribute to the initiation and progression of HF-PSF.

In patients with HF-PSF, the investigators will relate dietary changes to biochemical and cardiovascular functional measures. The investigators will study subjects on ad-lib diet and and following three weeks of rigorous dietary modification with the Dietary Approaches to Stop Hypertension (DASH)/sodium-restricted diet (SRD). This diet is richer in natural antioxidants and lower in sodium than the usual American diet. The DASH/SRD is recommended to lower blood pressure in patients with HTN, and is particularly effective in elderly, obese, and salt-sensitive hypertensives. Dietary sodium restriction is recommended for all HF patients including those with HF-PSF. The investigators hypothesize that the DASH/SRD will have favorable effects on oxidative stress, ventricular and vascular function, and blood pressure control in patients with hypertensive HF-PSF.

ELIGIBILITY:
Inclusion Criteria:

* Satisfy European Society of Cardiology guidelines for the diagnosis of HF-PSF (Paulus WJ et al. Eur. Heart J. 2007;28:2539-2550).
* Framingham criteria for heart failure satisfied
* left ventricular ejection fraction ≥ 50% (contrast ventriculography, echocardiography, nuclear scintigraphy)
* Diastolic dysfunction on previous echocardiogram/catheterization or evidence of abnormal neurohormonal activation (B-type natriuretic peptide (BNP) ≥ 100 pg/ml) with supporting evidence (atrial fibrillation, left atrial enlargement, left ventricular hypertrophy)
* History of systemic hypertension
* Willing to adhere to provided diet

Exclusion Criteria:

* New York Heart Association Class IV heart failure symptoms
* Hospitalization for decompensated heart failure within past one month
* Uncontrolled hypertension (seated systolic blood pressure ≥ 180 or diastolic blood pressure ≥ 110) at rest, on current antihypertensive regimen
* Changes in medical regimen for heart disease or hypertension within past 1 month, including diuretic dose adjustment
* Primary exercise limitation due to severe pulmonary disease
* Poor echocardiographic windows
* Worse than moderate mitral or aortic stenosis or insufficiency.
* Serum potassium level > 5.0 mmol/L at baseline or prior history of serum potassium level > 6.0
* Serum calcium/phosphorus product > 50 at baseline
* Severe renal insufficiency (current estimated glomerular filtration rate < 30 ml/min)
* Severe anemia (hemoglobin < 9 g/dL)
* Uncontrolled diabetes mellitus (hemoglobin A1c > 9%)
* Non-hypertensive cause of HF-PSF, e.g. amyloidosis, sarcoidosis, constrictive pericardial syndromes
* Myocardial infarction or unstable angina, including new or worsening anginal syndrome, within the past three months
* Uncontrolled arrhythmia (including non rate-controlled atrial fibrillation)
* Terminal illness expected to result in death within six months or active solid-organ cancer
* Psychiatric disorder or dementia with potential to compromise dietary adherence

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2009-07; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott L Hummel, MD MS, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

REFERENCES:
- [Background] Owan TE, Hodge DO, Herges RM, Jacobsen SJ, Roger VL, Redfield MM. Trends in prevalence and outcome of heart failure with preserved ejection fraction. N Engl J Med. 2006 Jul 20;355(3):251-9. doi: 10.1056/NEJMoa052256. PMID 16855265
- [Background] Redfield MM, Jacobsen SJ, Burnett JC Jr, Mahoney DW, Bailey KR, Rodeheffer RJ. Burden of systolic and diastolic ventricular dysfunction in the community: appreciating the scope of the heart failure epidemic. JAMA. 2003 Jan 8;289(2):194-202. doi: 10.1001/jama.289.2.194. PMID 12517230
- [Background] Klotz S, Hay I, Zhang G, Maurer M, Wang J, Burkhoff D. Development of heart failure in chronic hypertensive Dahl rats: focus on heart failure with preserved ejection fraction. Hypertension. 2006 May;47(5):901-11. doi: 10.1161/01.HYP.0000215579.81408.8e. Epub 2006 Apr 3. PMID 16585423
- [Background] Laffer CL, Bolterman RJ, Romero JC, Elijovich F. Effect of salt on isoprostanes in salt-sensitive essential hypertension. Hypertension. 2006 Mar;47(3):434-40. doi: 10.1161/01.HYP.0000202480.06735.82. Epub 2006 Jan 23. PMID 16432053
- [Background] Dekleva M, Celic V, Kostic N, Pencic B, Ivanovic AM, Caparevic Z. Left ventricular diastolic dysfunction is related to oxidative stress and exercise capacity in hypertensive patients with preserved systolic function. Cardiology. 2007;108(1):62-70. doi: 10.1159/000095883. Epub 2006 Sep 25. PMID 17003543
- [Background] Yugar-Toledo JC, Bonalume Tacito LH, Ferreira-Melo SE, Sousa W, Consolin-Colombo F, Irigoyen MC, Franchini K, Coelho OR, Moreno H Jr. Low-renin (volume dependent) mild-hypertensive patients have impaired flow-mediated and glyceryl-trinitrate stimulated vascular reactivity. Circ J. 2005 Nov;69(11):1380-5. doi: 10.1253/circj.69.1380. PMID 16247215
- [Background] Sacks FM, Svetkey LP, Vollmer WM, Appel LJ, Bray GA, Harsha D, Obarzanek E, Conlin PR, Miller ER 3rd, Simons-Morton DG, Karanja N, Lin PH; DASH-Sodium Collaborative Research Group. Effects on blood pressure of reduced dietary sodium and the Dietary Approaches to Stop Hypertension (DASH) diet. DASH-Sodium Collaborative Research Group. N Engl J Med. 2001 Jan 4;344(1):3-10. doi: 10.1056/NEJM200101043440101. PMID 11136953
- [Background] Paulus WJ, Tschope C, Sanderson JE, Rusconi C, Flachskampf FA, Rademakers FE, Marino P, Smiseth OA, De Keulenaer G, Leite-Moreira AF, Borbely A, Edes I, Handoko ML, Heymans S, Pezzali N, Pieske B, Dickstein K, Fraser AG, Brutsaert DL. How to diagnose diastolic heart failure: a consensus statement on the diagnosis of heart failure with normal left ventricular ejection fraction by the Heart Failure and Echocardiography Associations of the European Society of Cardiology. Eur Heart J. 2007 Oct;28(20):2539-50. doi: 10.1093/eurheartj/ehm037. Epub 2007 Apr 11. PMID 17428822
- [Result] Hummel SL, Seymour EM, Brook RD, Sheth SS, Ghosh E, Zhu S, Weder AB, Kovacs SJ, Kolias TJ. Low-sodium DASH diet improves diastolic function and ventricular-arterial coupling in hypertensive heart failure with preserved ejection fraction. Circ Heart Fail. 2013 Nov;6(6):1165-71. doi: 10.1161/CIRCHEARTFAILURE.113.000481. Epub 2013 Aug 28. PMID 23985432
- [Result] Hummel SL, Seymour EM, Brook RD, Kolias TJ, Sheth SS, Rosenblum HR, Wells JM, Weder AB. Low-sodium dietary approaches to stop hypertension diet reduces blood pressure, arterial stiffness, and oxidative stress in hypertensive heart failure with preserved ejection fraction. Hypertension. 2012 Nov;60(5):1200-6. doi: 10.1161/HYPERTENSIONAHA.112.202705. Epub 2012 Oct 1. PMID 23033371
- [Result] Mathew AV, Seymour EM, Byun J, Pennathur S, Hummel SL. Altered Metabolic Profile With Sodium-Restricted Dietary Approaches to Stop Hypertension Diet in Hypertensive Heart Failure With Preserved Ejection Fraction. J Card Fail. 2015 Dec;21(12):963-7. doi: 10.1016/j.cardfail.2015.10.003. Epub 2015 Oct 20. PMID 26497755
- See also: Hypertension publication from this study — http://www.ncbi.nlm.nih.gov/pubmed/23033371

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 22 patients screened, 14 enrolled
Groups:
- Dietary Intervention: Diet patterned after the intervention in the DASH-Sodium trial (Sacks FM et al. New Engl J Med 2001;344(1):3-10). The diet includes higher quantities of fresh fruits and vegetables, whole grain products, and low-fat dairy products than the standard American diet. The target sodium content is 50 mmol per 2100 kcal, and the caloric content is intended to maintain body weight. The diet is designed, prepared, and packaged by research dietitians and all food and beverages are provided for study participants.
  DASH/sodium-restricted diet (SRD) : Baseline diet will be assessed via Block Food Frequency Questionnaire, and 24-hour urinary sodium, potassium, and 8-isoprostanes will be measured. Subjects will then be assigned to 21 days of the DASH/SRD, with all food and beverages provided. Adherence will be assessed through a three-day food diary at the midpoint of the intervention, and at the end of the study urinary sodium, potassium, and 8-isoprostanes will again be measured.
Period: Overall Study
Arm/Group | Dietary Intervention
Started | 14
Completed | 13
Not Completed | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | Dietary Intervention
Number analyzed (Participants) | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 72 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 1
Region of Enrollment [Number; unit: participants]
  United States | 14
Body mass index [Mean (Standard Deviation); unit: kg/m^2] | 35.5 (7.9)
Hypertension [Count of Participants; unit: Participants] | 14
Participants with Chronic Kidney Disease [Count of Participants; unit: Participants] | 14
Coronary Artery Disease [Count of Participants; unit: Participants] | 5
Participants wtih Diabetes Mellitus [Count of Participants; unit: Participants] | 6
Participants wtih Anemia [Count of Participants; unit: Participants] | 6
New York Heart Assocation Classification [Count of Participants; unit: Participants] — NYHA class:
  I No limitation of physical activity. Ordinary physical activity does not cause undue fatigue, palpitation, dyspnea (shortness of breath).
  II Slight limitation of physical activity. Comfortable at rest. Ordinary physical activity results in fatigue, palpitation, dyspnea
  III Marked limitation of physical activity. Comfortable at rest. Less than ordinary activity causes fatigue, palpitation, or dyspnea.
  IV Unable to carry on any physical activity without discomfort. Symptoms of heart failure at rest. If any physical activity is undertaken, discomfort increases.
  Participants
    NYHA Class III | 12
    NYHA Class II | 2
Participants with prior hospitalization due to heart failure [Count of Participants; unit: Participants] | 10
Participants on chronic loop diuretics [Count of Participants; unit: Participants] | 11
Participants on 3 or more antihypertensive medications [Count of Participants; unit: Participants] | 10

OUTCOME MEASURES:

1. Primary Outcome: Brachial Artery Flow-mediated Dilation (FMD)
Time Frame: Prior to and following 21 days of dietary intervention, i.e. day 1 and day 22 of participation
Measure: Mean (Standard Deviation); unit: % dilation
Groups:
- Pre-dietary Intervention: Diet patterned after the intervention in the DASH-Sodium trial (Sacks FM et al. New Engl J Med 2001;344(1):3-10). The diet includes higher quantities of fresh fruits and vegetables, whole grain products, and low-fat dairy products than the standard American diet. The target sodium content is 50 mmol per 2100 kcal, and the caloric content is intended to maintain body weight. The diet is designed, prepared, and packaged by research dietitians and all food and beverages are provided for study participants.
  DASH/sodium-restricted diet (SRD) : Baseline diet will be assessed via Block Food Frequency Questionnaire, and 24-hour urinary sodium, potassium, and 8-isoprostanes will be measured. Subjects will then be assigned to 21 days of the DASH/SRD, with all food and beverages provided. Adherence will be assessed through a three-day food diary at the midpoint of the intervention, and at the end of the study urinary sodium, potassium, and 8-isoprostanes will again be measured.
Arm/Group | Pre-dietary Intervention | Post-dietary Intervention
Number analyzed (Participants) | 13 | 13
% dilation | 5 (5) | 8 (6)
Statistical Analysis 1: Comparison: Pre-dietary Intervention vs Post-dietary Intervention; Test type: Superiority or Other; p = .17, Wilcoxon matched-pairs

2. Secondary Outcome: Mean 24-hour Systolic Blood Pressure
Description: Change in 24-hour systolic blood pressure
Time Frame: Prior to and following 21 days of dietary intervention, i.e. day 1 and day 22 of participation
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Pre-dietary Intervention | Post-dietary Intervention
Number analyzed (Participants) | 13 | 13
mm Hg | 130 (4) | 123 (4)
Statistical Analysis 1: Comparison: Pre-dietary Intervention vs Post-dietary Intervention; Test type: Superiority or Other; p = .02, Wilcoxon matched-pairs tests

3. Secondary Outcome: Diurnal Variation in Ambulatory Blood Pressure
Description: Number of participants with non-dipping of nocturnal blood pressure - nighttime-to-daytime systolic BP ratio of >= 0.9
Time Frame: Prior to and following 21 days of dietary intervention, i.e. day 1 and day 22 of participation
Measure: Count of Participants; unit: Participants
Groups:
- Pre-Dietary Intervention: Diet patterned after the intervention in the DASH-Sodium trial (Sacks FM et al. New Engl J Med 2001;344(1):3-10). The diet includes higher quantities of fresh fruits and vegetables, whole grain products, and low-fat dairy products than the standard American diet. The target sodium content is 50 mmol per 2100 kcal, and the caloric content is intended to maintain body weight. The diet is designed, prepared, and packaged by research dietitians and all food and beverages are provided for study participants.
  DASH/sodium-restricted diet (SRD): Baseline diet will be assessed via Block Food Frequency Questionnaire, and 24-hour urinary sodium, potassium, and 8-isoprostanes will be measured. Subjects will then be assigned to 21 days of the DASH/SRD, with all food and beverages provided. Adherence will be assessed through a three-day food diary at the midpoint of the intervention, and at the end of the study urinary sodium, potassium, and 8-isoprostanes will again be measured.
- Post-dietary Intervention: Post-dietary intervention
Arm/Group | Pre-Dietary Intervention | Post-dietary Intervention
Number analyzed (Participants) | 13 | 13
Participants | 10 | 7

4. Secondary Outcome: Aortic Augmentation Index
Description: Aortic augmentation index is the ratio of the augmentation pressure to the central pulse pressure, expressed as a percentage. Both parameters are obtained via mathematical transformation of the radial pulse wave. The augmentation pressure represents the contribution of reflected waves to the pulse pressure. The central pulse pressure is the ratio between maximum aortic systolic pressure and minimum aortic diastolic pressure. A higher aortic augmentation index and central pulse pressure reflect increased arterial stiffness. Increased arterial stiffness is associated with an increased long-term risk of cardiovascular disease.
Time Frame: Prior to and following 21 days of dietary intervention, i.e. day 1 and day 22 of participation
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Pre-Dietary Intervention | Post-dietary Intervention
Number analyzed (Participants) | 12 | 12
percentage | 29 (9) | 28 (10)

5. Secondary Outcome: Carotid-femoral Pulse Wave Velocity
Time Frame: Prior to and following 21 days of dietary intervention, i.e. day 1 and day 22 of participation
Measure: Mean (Standard Deviation); unit: m/s
Arm/Group | Pre-Dietary Intervention | Post-Dietary Intervention
Number analyzed (Participants) | 11 | 11
m/s | 12.4 (3) | 11.0 (2.2)

6. Secondary Outcome: Ventricular Diastolic Function
Description: Lateral mitral annulus E/e' ratio
Time Frame: Prior to and following 21 days of dietary intervention, i.e. day 1 and day 22 of participation
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Pre-Dietary Intervention | Post-Dietary Intervention
Number analyzed (Participants) | 12 | 12
ratio | 12 (2) | 11 (2)

7. Secondary Outcome: Six Minute Walk Test Distance
Time Frame: Prior to and following 21 days of dietary intervention, i.e. day 1 and day 22 of participation
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Pre-Dietary Intervention | Post-Dietary Intervention
Number analyzed (Participants) | 13 | 13
meters | 313 (86) | 337 (91)
Statistical Analysis 1: Comparison: Pre-Dietary Intervention vs Post-Dietary Intervention; Test type: Superiority; p = .006, t-test, 2 sided

8. Secondary Outcome: Urinary 8-isoprostanes
Time Frame: Prior to and following 21 days of dietary intervention, i.e. day 1 and day 22 of participation
Measure: Mean (Standard Deviation); unit: mmol F2-iso/mmol Cr
Arm/Group | Pre-Dietary Intervention | Post-Dietary Intervention
Number analyzed (Participants) | 13 | 13
mmol F2-iso/mmol Cr | 70 (28) | 48 (15)
Statistical Analysis 1: Comparison: Pre-Dietary Intervention vs Post-Dietary Intervention; Test type: Superiority; p = .02, t-test, 2 sided

9. Other Pre Specified Outcome: EndoPAT Arterial Endothelial Function
Time Frame: Prior to and following 21 days of dietary intervention, i.e. day 1 and day 22 of participation
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Estimated Glomerular Filtration Rate, Serum Potassium, Serum Calcium-phosphorus Product
Description: Safety measures to determine adverse effects of the provided DASH diet home-delivered meals
Time Frame: Prior to and following 21 days of dietary intervention, i.e. day 1 and day 22 of participation
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 25 days
Arm/Group | Dietary Intervention
Serious Adverse Events (participants affected / at risk) | 0/14
Other Adverse Events (participants affected / at risk) | 1/14
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dietary Intervention (N=14)
hyperkalemia (Metabolism and nutrition disorders) | 1 (1) — At day 5 safety visit 1 subject had serum potassium 5.9, an expected potential adverse event in this protocol. There were no associated symptoms or sequelae, and the patient was withdrawn form the study diet as per protocol.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No